CLINICAL TRIAL: NCT03912454
Title: A Prospective Study of Clinical Outcomes Following a Single Intradiscal Injection of Bone Marrow Aspirate Concentrate (BMAC) for Single Level Discogenic Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bone and Joint Clinic of Baton Rouge (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMAC1601
Record Dates: First submitted 2019-04-10; First posted 2019-04-11 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Degenerative Disc Disease; Spine Degeneration
MeSH Terms: conditions — Intervertebral Disc Degeneration | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BMAC Injection (Experimental)
  Interventions: Other: Autologous Bone Marrow Aspirate Concentrate (BMAC) Injection

INTERVENTIONS:
Other: Autologous Bone Marrow Aspirate Concentrate (BMAC) Injection — Subjects will undergo bone marrow aspiration from the iliac crest. Bone marrow will be concentrated and injected into the symptomatic lumbar disc.

SUMMARY:
This single-institution prospective case series (single arm) study will assess the clinical outcomes of patients diagnosed with 1 or 2 level level discogenic low back pain following an intradiscal injection of bone marrow aspirate concentrate (BMAC).

DETAILED DESCRIPTION:
Background:

BMAC is a cellular rich fraction of bone marrow aspirate that can be readily prepared at the point of care without additional processing steps to manipulate or isolate cells. In addition, BMAC contains growth factors from the peripheral blood which may promote disc healing.

Study Summary:

The study population will consist of up to 20 patients aged 18- 60 with unresolved low back pain attributable to intervertebral disc degeneration. Clinical exam will indicate the intervertebral disc as the source of pain with features such as midline pain, pain upon rising from a seated position, or positive responses to centralization maneuvers. Moderate single level lumbar disc (L1-S1) degeneration (<50% disc height) will be confirmed on MRI. Other low back pain generators must be eliminated prior to study enrollment. Subjects must meet minimum score criteria on baseline PROs (VAS>=40 and ODI>=30). Subjects that meet all of the inclusion and none of the exclusion criteria will be invited to participate in the study.

Enrolled subjects will undergo bone marrow aspiration and intradiscal injection by an experienced orthopedic spine surgeon. Subjects will be followed for 1 year to evaluate the effects of the disc injection.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 to 60 years
* Symptomatic discogenic low back pain, clinically demonstrated by a loss of lumbar range of motion and pain to deep palpation over the symptomatic disc.
* MRI confirmed single level lumbar disc height loss <50% (Modified Pfirrman grade <=7).
* MRI confirmed isolated lumbar disc degeneration OR

  o If zygapophysial joint degeneration is present on MRI, subject must have failed intra-articular injection or medial branch block (<50% pain relief) to be eligible for enrollment. PI will have final discretion as to whether the patient's symptoms originate from a single disc.
* Patient must have completed at least 3 months conservative treatment. Conservative treatment may include NSAIDs or Acetaminophen when medically appropriate and physiotherapy, chiropractic care, or a guided home exercise program.
* BMI < 40
* Back pain greater than leg pain with back pain rating on a 100 mm visual analog scale (VAS) >= 40 mm
* Pain Catastrophizing Scale <= 30

Exclusion Criteria:

* Prior fusion at the level to be treated
* >2 levels requiring intervention
* Non discogenic source of back pain
* Intradural disc herniation
* Full thickness annular tear at the index level.
* Lumbar spine surgery within the past 6 months.
* Pregnant or breastfeeding.
* Known allergy or sensitivity to heparin or citrate (used for processing BMAC)
* Coagulopathy preventing spinal injection
* Active infection
* Malignancy within past 5 years other than basal cell or squamous cell skin cancer.
* Severe uncontrolled medical condition
* Other significant pain generator that may affect the subject's answers to PRO questionnaires.
* Current Tobacco use
* Pending litigation involving subject's back pain
* Incarcerated at the time of study enrollment
* Inability to give informed consent for study participation for any reason

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-04-08 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Change in Visual Analog Scale (VAS) Pain Score | 1 day (Pre-injection) to 12 months post-injection
  The severity of back and leg pain will be evaluated using a 100 mm visual analog scale (VAS) where a higher number indicates greater pain.
Change in Oswestry Disability Index | 1 day (Pre-injection) to 12 months post-injection
  The Oswestry Disability Index (ODI) is the most commonly used patient reported outcome measure in patients with low back pain. The ODI score ranges from 0% to 100%. A higher score corresponds to a greater disability.

SECONDARY OUTCOMES:
BMAC injection survival | 12 months post-injection
  The number of subjects who do not proceed to surgery for their discogenic back pain and answer YES to " Are you satisfied with the outcome of this injection? OR NO to "Are you seeking any additional treatments for your discogenic back pain at this time?"
MRI evaluation of the degenerative disc | 1 day (Pre-injection) and 12 months post-injection
  A modified Pfirrman grade will be assigned and used to assess changes in the disc pre-injection to 1 year post - injection
CFU-F Analysis | 1 Day of Injection
  Cell viability testing and CFU-F assay will be conducted on an aliquot from each subject's BMAC. Number of CFU-F from each patient will be used to correlate with patient reported outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Bone and Joint Clinic of Baton Rouge, Baton Rouge, Louisiana, United States